CLINICAL TRIAL: NCT00764010
Title: Diet and Omega-3 Intervention Trial on Atherosclerosis
Acronym: DOIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other); Ultrasound Laboratory at Malmoe University Hospital, Sweden (Other); Norwegian Retail Company RIMI (Unknown); Norwegian Cardiovascular Council (Unknown)
Responsible Party: Harald Arnesen, Professor of Medicine, Ulleval University Hospital, Oslo, Norway
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 175
Record Dates: First submitted 2008-09-26; First posted 2008-10-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Docosahexaenoic Acids; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): No dietary counseling, placebo capsules for omega-3
- 2 (Active Comparator): Dietary counseling, placebo capsules for omega-3
  Interventions: Dietary Supplement: Dietary counseling, placebo capsules for omega-3
- 3 (Active Comparator): No dietary counseling, omega-3 capsules
  Interventions: Dietary Supplement: No dietary counseling and omega-3 capsules
- 4 (Active Comparator): Dietary counseling and omega-3 capsules
  Interventions: Dietary Supplement: Omega-3 capsules and dietary counseling

INTERVENTIONS:
Dietary Supplement: No dietary counseling and omega-3 capsules — Omega-3 2.4 g/day
  Arms: 3
Dietary Supplement: Omega-3 capsules and dietary counseling — Omega-3 2.4 g/day and Mediterranean-like diet
  Arms: 4
Dietary Supplement: Dietary counseling, placebo capsules for omega-3 — Mediterranean-like diet
  Arms: 2

SUMMARY:
The study was actuated to evaluate the effects of a 3-year intervention with diet and/or very long chain omega-3 (VLC n-3 PUFA), in a randomized 2x2 factorial design on the progression of atherosclerosis in a high risk population. A total of 563 elderly men were included and randomized to receive usual care and VLC n-3 placebo capsules (control group), dietary advice and VLC n-3 placebo capsules, usual care and VLC n-3 capsules, and finally both VLC n-3 capsules and dietary advice.

The evaluation of atherosclerosis were i) ultrasound measurement of carotid intima media thickening ii) pulse wave propagation time iii) circulating biomarkers of atherosclerosis.

DETAILED DESCRIPTION:
The basis for recruitment was a follow up of subjects participating in the Oslo Diet and Anti Smoking Study (1972-1977) characterised as hypercholesterolemic in 1972.

Measurements of the outcome variables were performed at baseline and after 36 m; blood sampling also after 6 and 18 m.

In addition to the main outcome variables, a biobank was established for future analyses.

Clinical events were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elderly men with long standing hypercholesterolemia (cholesterol > 6.45 mmol/L and < 8.00 mmol/L) with or without coronary heart disease.

Exclusion Criteria:

* Cholesterol > 8.00 mmol/L, blood pressure > 170/100
* Uncontrolled hypertension
* Socially or otherwise unsuitable subjects
* Anticipated non compliance
* Other major non cardiac illness expected to reduce life expectancy or interfere with study participation.

Ages: 64 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 1997-05; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Variables of atherosclerosis progression: IMT, Pulse Wave Propagation Time, Circulating biomarkers | 1997-2010

SECONDARY OUTCOMES:
Genetical influence of the intervention principles ("Nutrigenetics") | 1997-2010

CONTACTS AND LOCATIONS:
Overall Officials: Harald Arnesen, M.D, PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ullevål University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Awoyemi A, Troseid M, Arnesen H, Solheim S, Seljeflot I. Markers of metabolic endotoxemia as related to metabolic syndrome in an elderly male population at high cardiovascular risk: a cross-sectional study. Diabetol Metab Syndr. 2018 Jul 21;10:59. doi: 10.1186/s13098-018-0360-3. eCollection 2018. PMID 30038669
- [Derived] Weiss TW, Arnesen H, Seljeflot I. Components of the interleukin-6 transsignalling system are associated with the metabolic syndrome, endothelial dysfunction and arterial stiffness. Metabolism. 2013 Jul;62(7):1008-13. doi: 10.1016/j.metabol.2013.01.019. Epub 2013 Feb 19. PMID 23428306
- [Derived] Einvik G, Ekeberg O, Klemsdal TO, Sandvik L, Hjerkinn EM. Physical distress is associated with cardiovascular events in a high risk population of elderly men. BMC Cardiovasc Disord. 2009 Mar 30;9:14. doi: 10.1186/1471-2261-9-14. PMID 19331677